CLINICAL TRIAL: NCT07378462
Title: A Retrospective Randomized Controlled Study Comparing Low-Level Laser Therapy and Ultrasound Therapy for Pain Reduction in Temporomandibular Disorders
Brief Title: A Retrospective Randomized Controlled Study Comparing the Effectiveness of Low-level Laser Therapy and Ultrasound Therapy in Reducing Pain and Increasing Maximum Mouth Opening in Forty-six Patients With Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Akunchan Shrestha, Senior Resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRC/2509/023
Record Dates: First submitted 2026-01-18; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Disorders (TMD); Temporomandibular Joint Disorder
Keywords: low-level laser therapy; Temporomandibular Disorder (TMD); ultrasound therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy; Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: An interventional, comparative, parallel-group clinical study conducted in patients diagnosed with temporomandibular disorders according to DC/TMD criteria. Participants were allocated into two groups to receive either Low-Level Laser Therapy or Therapeutic Ultrasound Therapy, and outcomes were assessed over five treatment sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-level laser therapy (Experimental): Participants in this arm received low-level laser therapy applied to the area of maximum pain in the temporomandibular region. The therapy was delivered using a single-probe laser emitting infrared radiation at a wavelength of 650 nm, with an energy density of 2 J/cm² and an output power of 80 mW for 3 minutes per session. Treatment was administered over five sessions.
  Interventions: Device: Low-Level Laser Therapy
- Ultrasound therapy (Experimental): Participants in this arm received therapeutic ultrasound applied to the affected temporomandibular region. Ultrasound was delivered at a frequency of 1 MHz and an intensity of 1.3 W/cm² in continuous mode for 5 minutes per side per session. Treatment was administered over five sessions.
  Interventions: Device: Ultrasound therapy

INTERVENTIONS:
Device: Low-Level Laser Therapy — Low-level laser therapy delivered using a single-probe laser emitting infrared radiation at 650 nm, with an energy density of 2 J/cm² and output power of 80 mW for 3 minutes per session, applied to the area of maximum pain.
  Other Names: Light Therapy, Low-Level; Photobiomodulation Therapy
  Arms: Low-level laser therapy
Device: Ultrasound therapy — Therapeutic ultrasound delivered at a frequency of 1 MHz and intensity of 1.3 W/cm² in continuous mode for 5 minutes per side per session, applied to the affected temporomandibular region.
  Other Names: Therapeutic ultrasound
  Arms: Ultrasound therapy

SUMMARY:
Temporomandibular disorders (TMDs) are the most common cause of non-dental orofacial pain, involving the temporomandibular joint (TMJ), masticatory muscles, or associated structures. Globally, TMD is the second most prevalent musculoskeletal pain condition after low back pain. Epidemiological data show a high prevalence of TMD symptoms, particularly among women and Asian populations, with significant disease burden reported in Nepal. Conservative management remains the mainstay of TMD treatment, as evidence supporting surgical intervention is limited and inconclusive.

Among conservative modalities, physical therapies such as ultrasound therapy and low-level laser therapy (LLLT) have gained attention for pain reduction and functional improvement. Ultrasound therapy produces thermal and non-thermal effects that enhance blood flow, reduce muscle spasm, improve tissue extensibility, and promote healing. LLLT, through photobiomodulation, acts at the cellular level by increasing ATP production, reducing inflammatory mediators, enhancing collagen synthesis, and providing analgesic and anti-inflammatory effects.

Although several international studies have evaluated ultrasound and LLLT individually or in combination, limited studies have directly compared their effectiveness in TMD, and no such studies have been conducted in Nepal. Therefore, this study aims to compare the effectiveness of therapeutic ultrasound and LLLT in reducing pain and improving mouth opening in patients with TMD presenting to BPKIHS.

This was a retrospective randomized controlled study conducted at the Department of Oral Medicine and Radiology, College of Dental Surgery, BPKIHS. A total of 46 patients diagnosed with myalgia of masticatory muscles and/or TMJ arthralgia according to DC/TMD criteria were included using purposive sampling. Patients were allocated into two groups: Group A received low-level laser therapy (650 nm wavelength, 2 J/cm² for 3 minutes) and Group B received therapeutic ultrasound (1 MHz, 1.3 W/cm², continuous mode for 5 minutes). Five treatment sessions had been administered over two weeks.

Pain intensity was assessed using the Visual Analogue Scale (VAS) at each visit, while inter-incisal mouth opening was measured using a metallic scale at baseline and at the final visit.

Primary outcome measure was the difference in VAS scores in patients undergoing ultrasound therapy and low-level laser therapy for temporomandibular disorder before and after therapy.

Secondary outcome measures included the difference in inter-incisal mouth opening before and after therapy and the effectiveness of ultrasound therapy and low-level laser therapy in reducing pain in patients with arthralgia and myalgia.

Data were analyzed using SPSS version 11.5. Descriptive statistics were calculated, and inferential tests including independent and paired t-tests (or non-parametric equivalents), ANOVA/Kruskal-Wallis tests, and logistic regression were applied where appropriate. Ethical clearance was obtained from the Institutional Review Committee, BPKIHS with Ref. 20/080/081-IRC, Code no. IRC/2509/023.

DETAILED DESCRIPTION:
INTRODUCTION Temporomandibular joint disorders (TMDs), the most common cause of pain of non-dental origin in the oro-facial region, comprise signs and symptoms involving the masticatory muscles, temporomandibular joint or both. The American Academy of Orofacial pain defines temporomandibular disorders (TMDs) as "a collective term that includes a number of clinical problems that involve the masticatory muscles, the Temporomandibular joint (TMJ) and the associated structures". Pain limiting mouth opening, asymmetrical jaw movements, and TMJ sounds are the most common findings in TMDs.

TMD is the 2nd most common musculoskeletal pain in world, with low back pain being the first. About 33% of the population has at least one TMD symptom and 3.6 to 7.0% of the population has TMD with sufficient severity that they desire treatment. Whereas the prevalence of TMD symptoms in Asian adolescents is found to be considerably higher reporting 61.4 % of population having one or more TMD symptom/s. Epidemiological study in Eastern part of Nepal showed TMDs affecting mostly women in the age group of 31-50 years with prevalence of more than 2/3rd among the total study samples.

TMJ pain is considered the most common cause of chronic orofacial pain that is excruciating in nature. There are different types of treatment for TMD. Conservative treatments for TMD include medication, physiotherapy, occlusal splints, self-management strategies, and interventions based on cognitive behavioral approaches. At present, a conservative treatment approach prevails over surgery, given it is less aggressive and usually results in satisfactory clinical outcomes in mild-moderate TMD. In fact, the evidence for the greatest effectiveness of surgical versus conservative intervention to reduce short-term pain in arthrogenic TMD is controversial and inconclusive.

Pharmaceutic therapies have been vastly used in the past 25 years to relieve the syndrome of TMD. The most effective pharmacological agents used to treat TMD include nonsteroidal anti-inflammatory drugs (NSAIDs), opioids, corticosteroids, anxiolytics, muscle relaxants, antidepressants, and anticonvulsants.

The various physical therapy methods used are moist heat, ultrasound, laser, exercises, transcutaneous electrical nerve stimulation (TENS), microwave, and manual therapy. These methods help in decreasing muscular spasms; treatment of contractures; relief and healing of sports-related injuries; relief of pain; increased extensibility and treatment of contractures for collagen tissue (scar tissue) and connective tissues; heating of joint structures; treatment to improve limited joint motion, decrease in joint stiffness, arthritis, peri-arthritis, and bursitis; wound healing and the healing of varicose ulcers.

Ultrasound heat therapy is one of the primary choices of treatment for TMD. The effects of ultrasound can be divided into thermal and non-thermal. Pulsed ultrasound at a low intensity causes non-thermal or mechanical effects known as acoustic streaming produced by the ultrasound beam within the tissue. Streaming is the unidirectional movement of tissue components exposed to the ultrasonic field primarily at the cell membrane interface. This effect is believed to influence cellular diffusion rates, membrane permeability, and nerve conduction and to accelerate synthesis of collagen. In short, non-thermal ultrasound is used for stimulation of tissue repair, reduction of edema, and treatment of trigger points for pain management.

While diagnostic imaging includes scanned beams operating from 1 to 50 MHz (up to intravascular imaging and high-frequency applications), a physical therapists use low frequency (0.75-3 MHz) to apply ultrasound to promote healing, loosen muscles and joints, relieve pain, and increase blood flow to stimulate natural body defenses.

Ultrasound is mainly applied by physical therapists who are trained to place the transducer using a coupling oil or gel over a muscular area with a moving rotary motion to minimize dwell time. The output is limited typically to a maximum of 3 watts/cm2. A continuous wave or pulsed mode is usually available, and a timer up to 10 min is usually required. In normal application, ultrasound can be applied near bones where additional heating can occur, including shear wave conversion, so the therapist must be vigilant, and keep the transducer moving, and keep asking if the patient feels excessive heat.

Therapeutic lasers have also had a wide benefit to patients. The core idea of all these non-surgical treatments is to lower the symptom intensity, thus improving the function of the maxilla-mandibular unit. Low-level laser therapy (LLLT) has recently been put under the spotlight, because the proponents claim its easy application, limited treatment time and minimum contraindication.

A light-based treatment that produces monochromatic and coherent light of a single wavelength is called low-level laser therapy (LLLT). It acts via photobiology or bio-stimulation, altering cell and tissue functions. It acts on the mitochondria, causing them to produce more adenosine triphosphate (ATP) and decrease cellular oxygen consumption. It increases serotonin and endorphin levels and decreases prostaglandin (PGE 2) and interleukin (IL-1) beta levels, thereby reducing pain. The inflammation is reduced by inhibiting plasminogen activator, which is responsible for collagen breakdown, and increases collagen deposition.

According to the DC/TMD classification, the different types of myalgia are fundamentally differentiated by their extension, though maintaining the general characteristics described. Local or localized myalgia (LM) is characterized by pain of muscular origin, but it is localized to the area of palpation on examination. In myofascial pain (MP), soreness and discomfort also originate in the muscle, as in myalgia, but extend to the limits of the considered muscle, beyond the area identified by palpation. Finally, referred myofascial pain (RP) is characterized by extension of the soreness and discomfort towards areas distant from the area identified in the examination and from the limits of the palpated muscle.

In our study, patients diagnosed with local myalgia of masticatory muscle and arthralgia of TMJ based on Diagnostic Criteria for Temporomandibular Disorders DC/TMD were selected as inclusion criteria. Despite its high prevalence, there is no general agreement concerning its treatment, as it often responds poorly to therapeutic approaches based on occlusion splints, physiotherapy, analgesia, anti-inflammatory, or muscle relaxants. Cases that are refractory to these conservative therapeutic approaches serve as the motivation to seek other treatments. Therefore, ultrasound heat therapy and Low-level laser therapy are included within the available therapeutic array in these refractory cases.

RATIONALE OF THE STUDY Ultrasonic therapy has shown to have a thermal mechanism achieved by a continuous frequency (100% duty cycle) and a non- thermal mechanism achieved by a pulsed frequency (50% duty cycle). Low Intensity Ultrasound (LIUS) therapy increases local metabolism, microcirculation, and also tissue regeneration along with extensibility of connective tissues. The mechanical energy released is transferred in the manner of acoustic compression waves, producing mechanical and thermal physiological changes in the targeted tissue. Thermal physiological changes refer to increasing the local tissue temperature, increasing the blood flow associated with the increasing of the flexibility and extensibility of tissue with diminished fluid viscosity.

Over the last decade, the interest in using laser photobiomodulation in reducing TMD pain and obtaining anti-inflammatory effects has increased. According to Karu (2001) Low Level Laser treatment is a non-thermal therapy which can promote cell and tissue alterations caused by different types of metabolic activation (increased vascularization and the formation of fibroblasts) which determines an increase in the recovery process and/or tissue healing with non-invasive characteristics.

To the best of our literature search, no studies had been carried out in our country regarding the use of therapeutic ultrasound and low-level laser therapy in temporomandibular disorders, despite the high incidence of this condition. This research therefore aimed to study the benefits of therapeutic ultrasound and low-level laser therapy in patients with temporomandibular disorders presenting to BPKIHS. The findings of this study, if favorable, could be proposed as an adjunctive treatment option for patients suffering from temporomandibular disorders.

OBJECTIVES The primary objective of this study was to compare the difference in pain intensity, measured using the Visual Analogue Scale (VAS), in patients with temporomandibular disorder who underwent ultrasound therapy and low-level laser therapy before and after treatment. The secondary objectives were to compare the change in inter-incisal mouth opening before and after therapy in patients treated with ultrasound therapy and low-level laser therapy, and to evaluate the comparative effectiveness of these two treatment modalities in reducing pain among patients diagnosed with arthralgia and myalgia.

MATERIALS AND METHODS This study is designed as a retrospective randomized controlled study and was conducted in the Department of Oral Medicine and Radiology, College of Dental Surgery, B. P. Koirala Institute of Health Sciences (BPKIHS). The study population comprised patients diagnosed with temporomandibular disorder attending the Department of Oral Medicine and Radiology at BPKIHS.

A purposive sampling technique was employed for sample selection. The expected sample size for the study was 46 participants. No separate control group was included in the study. The total duration of the study was one year. There were no conflicts of interest declared by the investigators. Ethical clearance was obtained from the Institutional Review Committee (IRC), BPKIHS (Reference No. 20/080/081-IRC, Code No. IRC/2509/023).

METHODS (INTERVENTION/PROCEDURE)

Clinical examination and therapeutic procedures were carried out using standard diagnostic and treatment instruments. These included sterile mouth mirrors, explorers, tweezers, surgical gloves, spirit swabs, and gauge pieces for routine clinical use. Pain assessment and measurement of inter-incisal mouth opening were performed using a metallic scale.

Therapeutic interventions were administered using an HMS ultrasound therapy machine for ultrasound therapy and an LX-16 Woodpecker laser machine for low-level laser therapy. Ultrasound gel was used as a coupling medium during ultrasound application. All instruments and equipment were used following standard infection control and clinical protocols.

FREQUENCY AND DURATION OF INTERVENTION/FOLLOW UP OF SUBJECTS

First visit:

Ultrasound therapy or Low-Level Laser Therapy (LLLT) was administered. Baseline parameters, including pain score and inter-incisal mouth opening, were recorded. The therapy duration was 5 minutes for ultrasound or 3 minutes for LLLT, with a total visit time of approximately 15 minutes.

Second visit:

Ultrasound therapy or LLLT was administered. Pain intensity was assessed using the Visual Analogue Scale (VAS). The therapy duration was 5 minutes for ultrasound or 3 minutes for LLLT, with approximately 2 minutes required for assessment.

Third visit:

Ultrasound therapy or LLLT was administered. VAS pain score was recorded. The therapy duration was 5 minutes for ultrasound or 3 minutes for LLLT, with approximately 2 minutes required for assessment.

Fourth visit:

Ultrasound therapy or LLLT was administered. VAS pain score was recorded. The therapy duration was 5 minutes for ultrasound or 3 minutes for LLLT, with approximately 2 minutes required for assessment.

Fifth visit:

Ultrasound therapy or LLLT was administered. Final evaluation of pain score and inter-incisal mouth opening was performed. The therapy duration was 5 minutes for ultrasound or 3 minutes for LLLT, with a total visit time of approximately 15 minutes.

PROCEDURES AND SCHEDULE The study was conducted on patients visiting the Department of Oral Medicine and Radiology, BPKIHS, Dharan, who were clinically diagnosed with temporomandibular disorders according to the DC/TMD criteria. The treatment protocol was explained to the patients, and written informed consent was obtained.

The selected patients were divided into two groups. Patients in Group A received low-level laser therapy, while patients in Group B received ultrasound therapy.

Group A - Low-Level Laser Therapy (LLLT):

A single-probe laser device generating infrared radiation of 650 nm wavelength was applied. The energy intensity at the most painful points in the affected area was adjusted to 3 J/cm² and applied for 3 minutes. The laser was applied at a distance of 2 mm. An LX 16 Woodpecker Laser unit was used.

Group B - Ultrasound Therapy:

Ultrasound therapy was performed at 1.3 W/cm² for 5 minutes per session per side. A coupling agent (ultrasound gel) was used as a lubricant. An INDOSONIC 102n ultrasound therapy machine was used at a frequency of 1 MHz in continuous mode. The pre-auricular skin over the affected TMJ was cleansed with sterile cotton soaked in 70% isopropyl alcohol before application. A thin layer of ultrasound gel was evenly spread over the transducer head, which was applied with light pressure and moved slowly in a continuous circular motion while maintaining full contact with the skin.

During the treatment period, participants were given all necessary temporomandibular disorder instructions known as Physical Self-Regulation (PSR).

At baseline and at the final visit, inter-incisal mouth opening was measured between the maxillary and mandibular central incisors using a metallic scale. During every follow-up visit, pain in the temporomandibular region was assessed using the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst pain).

The schedule and duration of treatment sessions followed a predefined protocol, details of which are provided separately. Participants who were not willing to continue with the treatment protocol at any stage were withdrawn from the study.

Stopping rules were applied to ensure appropriate clinical decision-making. Treatment was discontinued if there was no improvement in Visual Analogue Scale (VAS) scores after completion of five therapy sessions or if there was no improvement in inter-incisal mouth opening after five therapy sessions.

No adverse responses or side effects related to the therapeutic interventions were observed or considered relevant during the study period. There were no procedures or conditions for breaking treatment allocation codes, as none were applicable. Training and calibration of investigators were not required for the conduct of this study.

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data were entered into a Microsoft Excel spreadsheet and subsequently transferred to SPSS version 11.5 for statistical analysis. Coding was assigned for data entry. Monitoring of the study was carried out weekly by the guide and co-guides.

Statistical Methods

Descriptive analysis:

Mean, median, standard deviation, proportions, and interquartile range were calculated.

Inferential statistics:

Independent t-test or Mann-Whitney U test was applied to compare mean values between the two groups.

Paired t-test or Wilcoxon signed-rank test was applied to compare pre- and post-therapy values within the same group.

ANOVA or Kruskal-Wallis test was applied to compare more than two means. Logistic regression analysis was performed to assess the strength of association between dependent and independent variables.

CALCULATION OF SAMPLE SIZE:

Considering 95% confidence interval, 80% power of study and mean score of VAS score from the study of Khairnar, Sanyukta et al (2019). The sample size is estimated using the following formula:

N= [2 x (Zα/2 + Zβ)² x (S2)]/(µ1 - µ2)² S= S1 + S2/ 2

Where, Zα/2 =1.96 at 95% level of significance

Zβ = 0.84 at 80% power

S = Common standard deviation

S1= Standard deviation post treatment in Group A (LLLT)

S2= Standard deviation post treatment in Group B (Ultrasound Therapy)

μ₁ = Mean VAS score post treatment in Group A (LLLT)

μ2= Mean VAS score post treatment in Group B (Ultrasound Therapy)

Sample size, N = [2 x (1.96 + 0.84) ² x (1.62)] / (4.81 - 6.19) ² 40.5 / 1.9= 20.25 ~ 21 per group

With 10% of non-responsive rate in both groups, Expected sample size: 46

ANNEXURE I: Proforma

Patient's demographic details

Name:

Date:

Age:

OPD Number:

Sex:

Ph. No:

Marital status:

Socio-economic status:

Occupation:

Education:

Address:

Group: A / B Diagnosis: Arthralgia / Myalgia Side: Right / Left Visit 1st 2nd 3rd 4th 5th VAS score

Pain free mouth opening (mm):

Maximum unassisted opening (mm):

Maximum assisted opening (mm):

Group A: Low Level Laser therapy Group B: Ultrasound Therapy

ELIGIBILITY:
Inclusion Criteria:

- Patient diagnosed with myalgia of masseter and temporalis muscles and arthralgia of TMJ based on Diagnostic Criteria for Temporomandibular Disorders DC/TMD.

Exclusion Criteria:

* Patients who were not willing to participate in the research.
* Patients who were undergoing treatment or had already undergone treatment for temporomandibular disorders within the preceding three months.
* Patients who were taking antidepressants, analgesics, or antipsychotic medications.
* Patients who had structural bony abnormalities of the temporomandibular joint on radiographic examination.
* Patients with the presence of joint disorders.
* Pregnant women.
* Patients with a history of facial trauma or fractures of the facial bones.
* Patients who presented with severe pain.
* Patients with severely reduced mouth opening (i.e., less than 10 mm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Compare the difference in mean pain intensity scores in patients undergoing Low-Level Laser Therapy and Ultrasound Therapy for Temporomandibular Disorder before and after therapy. | From enrollment to the end of treatment at 2 weeks
  Description:
  Pain intensity was assessed using the Visual Analogue Scale (VAS). The VAS consisted of a 10-cm horizontal line, with the left end representing "no pain" (0) and the right end representing "worst imaginable pain" (10). Higher scores indicated greater pain intensity.
  Participants were instructed on the use of the scale and were asked to mark a single point on the line corresponding to their current level of temporomandibular joint pain. Pain scores were recorded at baseline (pre-therapy) and at subsequent visits during the treatment period. The change in pain intensity was calculated by comparing pre- and post-therapy scores and was expressed as percentage reduction in VAS score.

SECONDARY OUTCOMES:
Compare the difference in mean inter-incisal mouth opening in patients undergoing Low-Level Laser Therapy and Ultrasound Therapy for Temporomandibular Disorder pre- and post-therapy | From enrollment to the end of treatment at 2 weeks
  Maximum mouth opening was measured as the inter-incisal distance using a metallic scale. In dentate patients, the distance between the incisal edges of the maxillary and mandibular central incisors was measured at maximum voluntary mouth opening. In edentulous patients, the distance was measured between the crest of the maxillary and mandibular alveolar ridges at the midline. Measurements were recorded in millimeters.
Compare the effectiveness of Low-Level Laser Therapy and Ultrasound Therapy in reducing pain in patients with temporomandibular joint arthralgia and myalgia of the masseter and temporalis muscles. | From enrollment to the end of treatment at 2 weeks
  Pain intensity was assessed using the Visual Analogue Scale (VAS). The VAS consisted of a 10-cm horizontal line, with the left end representing "no pain" (0) and the right end representing "worst imaginable pain" (10). Higher scores indicated greater pain intensity.
  Participants were instructed to indicate a single point on the scale corresponding to their current pain level in the affected joint or muscle. Pain scores were recorded at baseline (pre-therapy) and after completion of therapy. The effectiveness of low-level laser therapy and ultrasound therapy was evaluated by comparing the change in VAS scores before and after treatment in patients diagnosed with arthralgia and myalgia.

CONTACTS AND LOCATIONS:
Locations (1):
- B.P. Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Yes
All Individual participant data (IPD) collected throughout the trial will be made available upon reasonable request. De-identified data from the 46 study participants will be shared with other researchers for academic and research purposes, subject to ethical approval and compliance with institutional policies and participant confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: All the data are collected and will be provided when and where required.

REFERENCES:
- [Background] Ramachandra, Vijayalakshmi & Mubeen, & Rajguru, Preeti. (2015). Phonophoresis in temporomandibular joint disorders: A clinical trial. Journal of Advanced Clinical & Research Insights. 2. 259-264. 10.15713/ins.jcri.90.
- [Background] Rai S, Ranjan V, Misra D, Panjwani S. Management of myofascial pain by therapeutic ultrasound and transcutaneous electrical nerve stimulation: A comparative study. Eur J Dent. 2016 Jan-Mar;10(1):46-53. doi: 10.4103/1305-7456.175680. PMID 27011739
- [Background] Cavalcanti MF, Silva UH, Leal-Junior EC, Lopes-Martins RA, Marcos RL, Pallotta RC, Diomede F, Trubiani O, De Isla N, Frigo L. Comparative Study of the Physiotherapeutic and Drug Protocol and Low-Level Laser Irradiation in the Treatment of Pain Associated with Temporomandibular Dysfunction. Photomed Laser Surg. 2016 Dec;34(12):652-656. doi: 10.1089/pho.2016.4195. Epub 2016 Nov 29. PMID 27898256
- [Background] Ren H, Liu J, Liu Y, Yu C, Bao G, Kang H. Comparative effectiveness of low-level laser therapy with different wavelengths and transcutaneous electric nerve stimulation in the treatment of pain caused by temporomandibular disorders: A systematic review and network meta-analysis. J Oral Rehabil. 2022 Feb;49(2):138-149. doi: 10.1111/joor.13230. Epub 2021 Aug 21. PMID 34289157
- [Background] Ahmad, Rehab & Mohamed Abd Elatief, Emad & Sayed, Wadida & Ali, Rania & Ashour, Essam & Abdelsamee, Mohamed. (2018). Effect of Conventional Therapy and Low-Level Laser Therapy on Pain and Limitations of Daily Functions in Patients with Temporomandibular Joint Dysfunction. International Journal of Physiotherapy and Research. 6. 2797-2805. 10.16965/ijpr.2018.154.
- [Background] Veijola M, Kellokumpu S, Rajaniemi H. The effect of varying doses of hCG on the in vivo uptake by rat testis and serum testosterone response. Horm Res. 1984;19(3):191-9. doi: 10.1159/000179887. PMID 6325320
- [Background] Panhóca, Vitor Hugo et al. "Increased Oral Health-Related Quality of Life Postsynergistic Treatment with Ultrasound and Photobiomodulation Therapy in Patients with Temporomandibular Disorders." Photobiomodulation, photomedicine, and laser surgery vol. 37, 11 (2019): 694-699. doi:10.1089/photob.2019.4697
- [Background] Khairnar, Sanyukta et al. "Comparative evaluation of low-level laser therapy and ultrasound heat therapy in reducing temporomandibular joint disorder pain." Journal of dental anesthesia and pain medicine vol. 19,5 (2019): 289-294.
- [Background] Lin YS, Huang MH, Chai CY. Effects of helium-neon laser on the mucopolysaccharide induction in experimental osteoarthritic cartilage. Osteoarthritis Cartilage. 2006 Apr;14(4):377-83. doi: 10.1016/j.joca.2005.10.010. Epub 2005 Dec 13. PMID 16359876
- [Background] Lin YS, Huang MH, Chai CY, Yang RC. Effects of helium-neon laser on levels of stress protein and arthritic histopathology in experimental osteoarthritis. Am J Phys Med Rehabil. 2004 Oct;83(10):758-65. doi: 10.1097/01.phm.0000137310.15943.19. PMID 15385784
- [Background] Carvalho CM, Lacerda JA, dos Santos Neto FP, de Castro IC, Ramos TA, de Lima FO, de Cerqueira Luz JG, Ramalho MJ, dos Santos JN, Pinheiro AL. Evaluation of laser phototherapy in the inflammatory process of the rat's TMJ induced by carrageenan. Photomed Laser Surg. 2011 Apr;29(4):245-54. doi: 10.1089/pho.2009.2685. PMID 21457090
- [Background] Sakurai Y, Yamaguchi M, Abiko Y. Inhibitory effect of low-level laser irradiation on LPS-stimulated prostaglandin E2 production and cyclooxygenase-2 in human gingival fibroblasts. Eur J Oral Sci. 2000 Feb;108(1):29-34. doi: 10.1034/j.1600-0722.2000.00783.x. PMID 10706474
- [Background] Bjordal JM, Couppe C, Chow RT, Tuner J, Ljunggren EA. A systematic review of low level laser therapy with location-specific doses for pain from chronic joint disorders. Aust J Physiother. 2003;49(2):107-16. doi: 10.1016/s0004-9514(14)60127-6. PMID 12775206
- [Background] Skinner SM, Gage JP, Wilce PA, Shaw RM. A preliminary study of the effects of laser radiation on collagen metabolism in cell culture. Aust Dent J. 1996 Jun;41(3):188-92. doi: 10.1111/j.1834-7819.1996.tb04854.x. PMID 8768644
- [Background] Chen, J et al. "Efficacy of low-level laser therapy in the treatment of TMDs: a meta-analysis of 14 randomised controlled trials." Journal of oral rehabilitation vol. 42,4 (2015): 291-9. doi:10.1111/joor.12258
- [Background] Allen LV, Popovich NG, Ansel HC. Ansel's pharmaceutical dosage forms and drug delivery systems. Transdermal Drug Delivery Systems. 8th ed. India: Gopsons Papers Ltd.; 2006. p. 298 315.
- [Background] Baker KG, Robertson VJ, Duck FA. A review of therapeutic ultrasound: biophysical effects. Phys Ther. 2001 Jul;81(7):1351-8. PMID 11444998
- [Background] 10. Szabo, T. L. (2004). ULTRASOUND-INDUCED BIOEFFECTS. Diagnostic Ultrasound Imaging, 489-516. doi:10.1016/b978-012680145-3/50016-5
- [Background] Draper DO. Facts and misfits in ultrasound therapy: steps to improve your treatment outcomes. Eur J Phys Rehabil Med. 2014 Apr;50(2):209-16. Epub 2014 Mar 5. PMID 24594854
- [Background] Shukla D, Muthusekhar MR. Efficacy of low-level laser therapy in temporomandibular disorders: A systematic review. Natl J Maxillofac Surg. 2016 Jan-Jun;7(1):62-66. doi: 10.4103/0975-5950.196127. PMID 28163481
- [Background] Rahimi A, Rabiei S, Mojahedi SM, Kosarieh E. Application of low level laser in temporomandibular disorders. J Lasers Med Sci 2011; 2: 165-70.
- [Background] Shivhare P, Singh V, Giri R, Singh A, Penumatcha MR, Taparia N, Sabah N. Prevalence of temporomandibular disorders among Nepalese population. Journal of Chitwan Medical College. 2019; 9(29):34-42
- [Background] Lei J, Fu J, Yap AU, Fu KY. Temporomandibular disorders symptoms in Asian adolescents and their association with sleep quality and psychological distress. Cranio. 2016 Jul;34(4):242-9. doi: 10.1179/2151090315Y.0000000021. Epub 2016 Apr 28. PMID 27125298
- [Background] Von Korff M, Dworkin SF, Le Resche L, Kruger A. An epidemiologic comparison of pain complaints. Pain. 1988 Feb;32(2):173-183. doi: 10.1016/0304-3959(88)90066-8. PMID 3362555
- [Background] Scrivani SJ, Keith DA, Kaban LB. Temporomandibular disorders. N Engl J Med. 2008 Dec 18;359(25):2693-705. doi: 10.1056/NEJMra0802472. No abstract available. PMID 19092154
- [Background] Mazzetto MO, Carrasco TG, Bidinelo EF, de Andrade Pizzo RC, Mazzetto RG. Low intensity laser application in temporomandibular disorders: a phase I double-blind study. Cranio. 2007 Jul;25(3):186-92. doi: 10.1179/crn.2007.029. PMID 17696035
- [Background] Carrasco TG, Mazzetto MO, Mazzetto RG, Mestriner W Jr. Low intensity laser therapy in temporomandibular disorder: a phase II double-blind study. Cranio. 2008 Oct;26(4):274-81. doi: 10.1179/crn.2008.037. PMID 19004308